CLINICAL TRIAL: NCT07003581
Title: Cardiometabolic Risk Factors Associated With Multidrug-Resistant Tuberculosis: A Case-Control Study
Brief Title: Cardiometabolic Risk Factors Associated With Multidrug-Resistant Tuberculosis
Status: Completed | Type: Observational
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Sishir Poudel, Doctor, B.P. Koirala Institute of Health Sciences
Other Study IDs: 441_2024
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Tuberculosis (TB)
Keywords: Tuberculosis; Multidrug resistant
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: MDR-TB patient
- Control: Drug sensitive TB patient

SUMMARY:
Background: MDR-TB (Multidrug Resistant tuberculosis) remains a major public health concern, especially in high-burden countries like Nepal. While individual risk factors are known, the cumulative impact of cardiometabolic on MDR-TB is not well understood.

Methods and Findings: A health-facility-based, age- and sex-matched 1:2 case-control study will be conducted at DR-TB (Drug Resistant Tuberculosis) treatment centers in Gandaki Province, Nepal. MDR-TB patients (cases) and DS-TB patients (controls) will be enrolled. Cases will be defined as adults (≥18 years) with confirmed MDR-TB; controls will be adults with sputum-positive DS-TB (Drug Sensitive Tuberculosis). Data on sociodemographics, cardiometabolic risk factors (alcohol, tobacco, BMI, hypertension, diabetes), TB literacy, and treatment history will be collected using a structured, pretested questionnaire by trained medical officers. Data will be analyzed using SPSS v25. Binary logistic regression will be used to assess associations between risk factors and MDR-TB. Ethical approval will be obtained from the NHRC, and written informed consent will be obtained from all participants.

DETAILED DESCRIPTION:
Materials and Methods Study Design and Setting A health-facility-based, age- and sex-matched 1:2 case-control study will be conducted from September 2024 to February 2025 at DR-TB treatment centers in Gandaki Province, Nepal. These centers will include the Tuberculosis Treatment Center (Pokhara), Madhyabindu District Hospital (Nawalpur), and Dhawalagiri Hospital (Baglung). These centers are specialized facilities providing comprehensive TB care and treatment services, including for drug-resistant tuberculosis (DR-TB). They serve diverse populations from urban, semi-urban, and rural areas, ensuring a representative sample of the region's TB patients. The selection of these centers will allow for broad geographical representation and access to a large number of DR-TB patients.

Cases and Controls Selection The study will include patients undergoing treatment at DR-TB treatment centers in Gandaki Province. Cases will consist of patients diagnosed with MDR-TB, while controls will be patients with drug-susceptible TB (DS-TB) who are also receiving treatment at the same centers. To ensure comparability, each MDR-TB case will be matched with one or more DS-TB controls based on key demographic variables such as age and gender.

Cases A participant will be eligible to be included as a case if they are aged 18 years or older and diagnosed with MDR-TB (resistant to at least rifampicin and isoniazid) for the first time at the time of enrollment.

Controls A participant will be eligible to be included as a control if they are aged 18 years or older, diagnosed with sputum smear-positive DS-TB for the first time, and have received at least two weeks of anti-TB treatment.

Matching Criteria

A hierarchical procedure will be used to match controls with cases using the following variables, in order of importance:

Sex

Same age ± 5 years

Measurements

The primary exposure variables will include five key cardiometabolic risk factors:

Alcohol use - defined as current or past habitual consumption of alcoholic beverages.

Tobacco use - current or past smoking or smokeless tobacco consumption.

Body Mass Index (BMI) - calculated from measured height and weight and categorized according to WHO standards: underweight (<18.5 kg/m²), normal (18.5-24.9 kg/m²), overweight (25.0-29.9 kg/m²), and obese (≥30 kg/m²).

Hypertension - based on prior diagnosis, current use of antihypertensive medications, or blood pressure ≥140/90 mmHg.

Diabetes Mellitus (DM) - identified by self-reported diagnosis, anti-diabetic treatment, or fasting blood glucose ≥126 mg/dL.

Participants will be grouped into two categories based on the presence of these risk factors:

At least one cardiometabolic risk factor

No cardiometabolic risk factors

Additional Background Variables

Additional covariates will include:

Sociodemographic Characteristics: Age, sex, ethnicity, place of residence (rural/urban), occupation, educational attainment, marital status, type of settlement (temporary/permanent), and household size.

TB Literacy: Participants' knowledge regarding tuberculosis will be evaluated using a structured questionnaire covering TB transmission, prevention methods, and treatment practices.

Disease-Specific Factors: These will include history of contact with a known TB case, prior TB diagnosis, number of TB episodes, history of TB treatment interruption (including interruptions ≥1 week), medication history, treatment outcomes from previous episodes (e.g., cured, failed), and presence of coexisting conditions such as HIV/AIDS.

Sample Size Determination and Recruitment The sample size will be calculated using Epi-Info 7.2 statistical software. The parameters will include a prevalence of previously treated TB among controls of 10.4%, an odds ratio for MDR-TB among previously treated patients of 2.8, a 1:2 case-to-control ratio, 90% power, and 95% confidence level.

To adjust for potential non-response, the initially calculated sample size of 146 will be increased by 10%, resulting in a total of 162 participants: 54 cases and 108 controls. All cases and controls who fulfill the inclusion criteria will be consecutively enrolled until the required sample size is achieved.

Sample size formula:

N = ((Z<sub>1-α/2</sub> + Z<sub>1-β</sub>)² × (p₀q₀ + p₁q₁)) / (p₁ - p₀)²

p₀ = likely proportion of previous treatment history among controls

q₀ = 1 - p₀

p₁ = likely proportion among cases

q₁ = 1 - p₁

α = significance level

1 - β = power of the test

Data Collection Tools and Study Procedures Data will be collected face-to-face using a structured, bilingual (English and Nepali), and pre-tested survey questionnaire adapted from existing literature. Patient recruitment will occur over a 16-week period, from 1st September 2024 to 31st December 2024. After obtaining written informed consent, each participant will be interviewed using a standardized questionnaire in their preferred language (English or Nepali). To minimize recall bias, a Nepali calendar will be used for referencing dates. Data will be collected using the KoboCollect app. All interviews will be conducted by trained medical officers.

Data Analysis Initially, the raw data will be entered into Microsoft Excel, where it will undergo cleaning and consistency checks. Descriptive statistics will be presented as means and standard deviations for continuous variables and frequencies and percentages for categorical variables. Multivariate logistic regression will be used to identify independent associations between cardiometabolic risk factors and MDR-TB, controlling for relevant background variables. Adjusted odds ratios (AORs) with 95% confidence intervals (CIs) will be reported. A p-value of less than 0.05 will be considered statistically significant. All statistical analyses will be performed using SPSS version 25 (IBM, Armonk, NY).

Ethical Considerations Ethical approval will be obtained from the Nepal Health Research Council. Permission will also be obtained from hospital administrations to approach participants for data collection (Protocol Registration No: 441_2024). Before data collection, the nature and purpose of the study will be explained to participants verbally, and written informed consent will be obtained. Participants' anonymity and confidentiality will be ensured throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Diagnosed with multidrug-resistant TB (MDR-TB) (resistant to at least isoniazid and rifampicin), confirmed by drug susceptibility testing or GeneXpert or Drug Sensitive TB
* Newly diagnosed with MDR-TB (i.e., not previously treated for MDR-TB) or DS-TB.
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Patients with extrapulmonary TB only, without confirmed pulmonary involvement.
* Patients with severe illness or comorbidities that preclude participation in an interview (e.g., unconscious, severely mentally ill).
* Pregnant women (if cardiometabolic variables like BMI or BP may be physiologically altered).
* Participants who refuse or are unable to provide informed consent.
* Patients who have incomplete or missing data on key exposure or outcome variables.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients undergoing treatment at drug-resistant tuberculosis (DR-TB) treatment centers in Gandaki Province. Cases will consist of patients diagnosed with MDR-TB while controls will be patients with drug-susceptible (DS-TB) who are also receiving treatment at the same centers. To ensure comparability, each MDR-TB case will be matched with one or more drug-susceptible TB controls based on key demographic variables such as age and gender.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Multidrug-Resistant Tuberculosis (MDR-TB) status | At the time of study enrollment (cross-sectional capture of TB drug resistance status at diagnosis)
  This outcome is assessed retrospectively based on confirmed laboratory diagnosis at the DR-TB treatment centers.

CONTACTS AND LOCATIONS:
Locations (1):
- Mustang Hospital, Jomsom, Nepal

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to the sensitive and confidential nature of tuberculosis-related information. Tuberculosis remains a highly stigmatized condition in many communities, including in Nepal, and sharing participant-level data could potentially compromise patient privacy and confidentiality, even if de-identified